CLINICAL TRIAL: NCT05066971
Title: Personalized Medicine: Home Monitoring as a Tool to Patient Empowerment. Rate Control Self-adjustment in Patients With Permanent or Persistent Atrial Fibrillation Using Cardiovascular Implantable Electronic Device (CIED) Information
Brief Title: Rate Control Self-adjustment in Patients With Permanent or Persistent Atrial Fibrillation Using Device Home Monitoring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Félix Ayala-Paredes, Cardiologist, electrophysiologist, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-2913
Record Dates: First submitted 2021-06-12; First posted 2021-10-04 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation, Persistent
Keywords: Atrial fibrillation; Patient empowerment; Personalized medicine; Rate control
MeSH Terms: conditions — Atrial Fibrillation; Patient Participation

STUDY DESIGN:
Intervention Model Description: All participants follow the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants in gradual self-adjustment rate control medication (Experimental): Patients receive a weekly simplified version of the information transmitted by the HM system. In the first 3 months, using that information, the physician changes or not the rate control medication posology (i.e. if the mean heart rate is 60bpm, betablocker dose is cut to half, and another heart rate evaluation is done a week later, and if heart rate is now 120bpm the dose is increased to a 3/4 of the initial dose, and so on). After those three initial months where physician guide titration, the patient is allowed to make self-adjustment of their medication accordingly to the information received (i.e. increasing or decreasing their rate control medication depending on heart rates and activity hours per day.
  Interventions: Combination Product: Self-adjustment of medication

INTERVENTIONS:
Combination Product: Self-adjustment of medication — Each week, based on the information provided by HM (heart rate and hours of activity each day), the rate control medication is adjusted to increase the total of activity time.

SUMMARY:
Patients with permanent or persistent atrial fibrillation require rate control medication to prevent excessive tachycardia. Since too much medication leads to a lower than expected heart rate (low output and symptoms) and too little leads to a fast heart rate (with associated symptoms), finding the ideal medication level (target that could fluctuate) is vital for patient's wellbeing. Clinicians adjust the medication each time patients come into the clinic (once or twice a year). In between those visits, medication is not changed even though patients would benefit for some incremental medication adjustment.

Patients implanted with Biotronik devices have access to Home Monitoring® (HM), a user friendly remote monitoring system transmitting daily device and patient information to clinicians. Heart rate and activity hours can be tracked and this information could be used to adjust medication.

In a step by step process, patients will gradually gain autonomy in the weekly adjustment of their rate control medication. In order to guide medication adjustment by patients, the research team will filter and simplify the information received by HM before sending it to patients. It is hypothesize that patient empowerment, understanding the dynamics of their heart rates in relation to the amount of medication used, will lead to better heart rate control, and it will improve the daily hours of patients activity.

DETAILED DESCRIPTION:
Patients with permanent or persistent atrial fibrillation require rate control medication to prevent heart rate (HR) speed up. Beta-blockers or calcium channel blockers are used to achieve a reasonable HR; symptoms, EKG and Holter recordings guide clinicians to rate control targets at clinical encounters (at our pacemaker clinic at 6 to 12 months intervals). Once a target HR is achieved, unless new symptoms arise, medication is seldom modified. Rate control medications need to be well adjusted: if not enough dose administered, HR will increase, leading to palpitations, shortness of breath and eventually heart failure; if too much medication is given, patients would experience low cardiac output symptoms (fatigue, tiredness, shortness of breath, low blood pressure, and eventually syncope). Clinicians tend to over control heart rates with no added benefits.

Most of patients with a pacemaker or defibrillator at our center are offered a remote monitoring system as part of a regular follow up schema at our pacemaker clinic; usually to reduce in face encounters, and to be alerted if a problem arises with the pacemaker or defibrillator. There are many remote monitoring systems (five, one for each vendor implanted at our center), and the Home Monitoring® (HM) from Biotronik is specially friendly as all information from the device (pacemaker or defibrillator) is transmitted every day to our clinic with no interaction from the patient side. Beside device status itself (remaining battery, system integrity) daily mean heart rates (measured in beats per minute: bpm) and patient activity (measured as hours per day in activity, as detected by the movement or activity sensor implanted in the device) are also transmitted, but if HR are between safety boundaries (programmed for each patient after implant), all information is rarely used for any other purpose.

If patients with permanent or persistent atrial fibrillation, rate control stable medication, and a HM pacemaker, are followed closely (every week) to adjust the medication (every week if needed, by the research team at the beginning) based on mean heart rates and daily activities already received, we hypothesize that patients will achieve not only better rate control targets, but they will increase their hours of activity per day. Eventually once the patient has understood the principle, medication adjustment would be done by the patient itself based on the same simple information redirected to him or her.

ELIGIBILITY:
Inclusion Criteria:

* patients with persistent or permanent atrial fibrillation, on rate control medication stable for at least 6 months
* patients with a Biotronik pacemaker connected to HM system

Exclusion Criteria:

* patients with heart failure in need of maximum beta blocker titration
* patients with other indications that would prevent medication adjustment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
6 minutes walk test | Baseline, end of the study (12 months after first 6 minute walk test)
  Difference in meters walked between first and last 6 minutes walk test
Heart rate control target | Through study completion, up to 1 year
  Number of weeks where the heart rate is between 80 and 110 beats per minute
Physical activity during the day | Through study completion, up to 1 year
  Percentage of physical activity during the day measured by the pacemaker accelerometer at the end of each week

CONTACTS AND LOCATIONS:
Overall Officials: Felix Alejandro Ayala Paredes, MD PhD, Principal Investigator — Sherbrooke university medical school
Locations (1):
- CHUS Fleurimont, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Gelder IC, Groenveld HF, Crijns HJ, Tuininga YS, Tijssen JG, Alings AM, Hillege HL, Bergsma-Kadijk JA, Cornel JH, Kamp O, Tukkie R, Bosker HA, Van Veldhuisen DJ, Van den Berg MP; RACE II Investigators. Lenient versus strict rate control in patients with atrial fibrillation. N Engl J Med. 2010 Apr 15;362(15):1363-73. doi: 10.1056/NEJMoa1001337. Epub 2010 Mar 15. PMID 20231232
- [Background] Yee R, Verma A, Beardsall M, Fraser J, Philippon F, Exner DV. Canadian Cardiovascular Society/Canadian Heart Rhythm Society joint position statement on the use of remote monitoring for cardiovascular implantable electronic device follow-up. Can J Cardiol. 2013 Jun;29(6):644-51. doi: 10.1016/j.cjca.2012.11.036. Epub 2013 Mar 5. PMID 23465345
- [Background] Chronaki CE, Vardas P. Remote monitoring costs, benefits, and reimbursement: a European perspective. Europace. 2013 Jun;15 Suppl 1:i59-i64. doi: 10.1093/europace/eut110. PMID 23737233
- [Background] Slotwiner D, Varma N, Akar JG, Annas G, Beardsall M, Fogel RI, Galizio NO, Glotzer TV, Leahy RA, Love CJ, McLean RC, Mittal S, Morichelli L, Patton KK, Raitt MH, Ricci RP, Rickard J, Schoenfeld MH, Serwer GA, Shea J, Varosy P, Verma A, Yu CM. HRS Expert Consensus Statement on remote interrogation and monitoring for cardiovascular implantable electronic devices. Heart Rhythm. 2015 Jul;12(7):e69-100. doi: 10.1016/j.hrthm.2015.05.008. Epub 2015 May 14. No abstract available. PMID 25981148